CLINICAL TRIAL: NCT04071288
Title: Comparison of Burch Colposuspension and Mid-urethral Sling Operations for Stress Urinary Incontinence
Brief Title: Burch Colposuspension and Mid-urethral Sling Operations
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, pınar kadiroğulları M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2018.02.02
Record Dates: First submitted 2019-08-24; First posted 2019-08-28 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laparoscopic burch colposuspension: who underwent total laparoscopic hysterectomy for benign causes and had simultaneous incontinence; patients undergoing laparoscopic burch colposuspension
  Interventions: Procedure: total laparoscopic hysterectomy and simultaneous incontinence surgery with benign causes
- mid urethral sling operations: who underwent total laparoscopic hysterectomy for benign causes and had simultaneous incontinence; patients undergoing mid-urethral sling operations
  Interventions: Procedure: total laparoscopic hysterectomy and simultaneous incontinence surgery with benign causes

INTERVENTIONS:
Procedure: total laparoscopic hysterectomy and simultaneous incontinence surgery with benign causes — total laparoscopic hysterectomy and simultaneous incontinence surgery with benign causes; Burch colposuspension and mid-urethral sling operations for stress urinary incontinence

SUMMARY:
Stress urinary incontinence is common in women. the treatment of this condition is surgery. investigators add stress incontinence surgery to patients who undergo total laparoscopic hysterectomy for benign reasons.

Depending on the patient's general condition and indications, the operation can be performed by vaginal approach, as well as mid-urethral sling operations and laparoscopic burch colposuspension.

The researchers aimed to compare these two types of operations performed on patients. In this way, the superiority and disadvantage of each other in two procedures will be demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* A total laparoscopic hysterectomy was planned for benign causes,
* Patients scheduled for simultaneous operation for incontinence

Exclusion Criteria:

* Patients previously operated for urinary incontinence
* Patients whose diagnosis of stress urinary incontinence is uncertain
* Patients with urinary tract infection

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total laparoscopic hysterectomy was planned for benign causes, Patients who underwent simultaneous operation for incontinence
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
recurrence | 2 years
  in patients who underwent total laparoscopic hysterectomy and simultaneous incontinence surgery for benign reasons; In the early postoperative period, relapse will be evaluated at 1 month, 6 months and 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)